CLINICAL TRIAL: NCT00759122
Title: EEG Biomarkers of Response in Depression
Brief Title: Electroencephalography (EEG) Biomarkers of Response in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Medtronic - MITG (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Ian A. Cook, MD, UCLA Semel Institute for Neuroscience and Human Behavior
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Biomarkers in MDD
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Major Depressive Disorder
Keywords: mdd; major depressive disorder; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): VENLAFAXINE
  Interventions: Drug: venlafaxine (Effexor)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: venlafaxine (Effexor) — Matching capsules containing venlafaxine 37.5 mg. WERE prepared by the UCLA Pharmacy for the initial phase of the study. After a one-week placebo lead-in, subjects WERE randomly assigned to receive one capsule of either venlafaxine or placebo, with the dosage increase every two days until subjects received four capsules daily (subjects achieved a dose of 150 mg. of venlafaxine after 10 days). The first dose was administered in the morning, with subsequent capsules added on a b.i.d. schedule.
  Arms: 1
Drug: placebo — Matching capsules containing placebo 37.5 mg. WERE prepared by the UCLA Pharmacy for the initial phase of the study. After a one-week placebo lead-in, subjects WERE randomly assigned to receive one capsule of either venlafaxine or placebo, with the dosage increase every two days until subjects received four capsules daily (subjects achieved a dose of 150 mg. of venlafaxine after 10 days). The first dose was administered in the morning, with subsequent capsules added on a b.i.d. schedule.
  Arms: 2

SUMMARY:
There are two specific aims of this project:

1. To identify physiologic indicators of venlafaxine treatment response using quantitative EEG (QEEG) cordance, and to determine if cordance changes are specifically associated with response to venlafaxine
2. To identify predictors of placebo response in major depression using QEEG cordance/bispectral index (BIS) and neuropsychological testing

DETAILED DESCRIPTION:
Our previous work indicates that a combination of neurophysiologic, symptom, and cognitive measures may predict response more accurately than brain functional measures alone. The purpose of this study is to replicate results from our earlier work using a similar study design (96-06-291-11), and also to prospectively gather additional information to substantiate that a more comprehensive approach to subject assessment will yield more accurate and reproducible prediction of treatment response.

One of the major challenges involved in clinical trials for major depressive disorder (MDD) is that of placebo response. The placebo response rate has been estimated at 20 - 50% of those subjects who enter a standard clinical trial for MDD. This high rate of response to placebo, which may not differ substantially from the response rate to medication, can make it difficult to demonstrate the efficacy of new antidepressant compounds. Identification of MDD subjects with a placebo responder (PR) phenotype, either at the beginning or end of a clinical trial, could have two major potential benefits. First, identification of placebo responders prior to enrollment in a clinical trial might make it possible to have restrictive entry criteria, excluding such subjects from the trial. Segregation of PR phenotype subjects a priori could reduce variance in the outcome data and increase the drug-placebo difference. This exclusion could reduce the number of subjects required for clinical trials and render the trials more efficient. Second, identification of a PR phenotype during a clinical trial could make it possible to distinguish "true medication" from placebo response. This distinction could make it possible to identify subgroups in the trial, enhancing precision in the study of medication effects.

Our research group has performed a series of placebo-controlled treatment trials in MDD and has used a combination of behavioral ratings, self-report, and neurophysiologic measurements with quantitative electroencephalography (QEEG) to identify predictors of both placebo response and medication response. The preliminary results from previous studies suggest that a combination of neurophysiologic, symptom, and cognitive measures may be useful for pretreatment prediction and/or early treatment detection of different types of treatment response.

In this study our primary goal is to assess the neurophysiologic, behavioral, and cognitive assessments of subjects with MDD in the setting of a clinical trial to replicate prospectively these initial results and more completely identify the characteristics of different types of treatment response in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will meet DSM-IV criteria for depression on the basis of a SCID-P interview, with subjects having a score on the 17-item Ham-D > 17 (with item #1 > 2).
* Subjects will meet criteria both at recruitment and after a one-week single blind placebo wash-in. Study includes outpatients only.

Exclusion Criteria:

* All subjects will have no serious medical illness. The investigators will exclude patients also meeting criteria for the following groups of axis I diagnoses:

  * delirium or dementia
  * substance-related disorders
  * schizophrenia or other psychotic disorders, or eating disorders.
* In addition, patients meeting criteria for cluster A or B axis II diagnoses will be excluded.
* Subjects with a history of current or past active suicidal ideation, or suicide attempts will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-11; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, MD, Principal Investigator — Professor
Locations (1):
- UCLA Laboratory of Brain, Behavior, and Pharmacology, Los Angeles, California, United States